CLINICAL TRIAL: NCT04257669
Title: The Relationship Between Iron Status, Cognitive Performance, Subjective Mood and Fatigue in Women of Reproductive Age
Status: Completed | Type: Observational
Sponsor: Northumbria University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 9BM1
Record Dates: First submitted 2020-01-29; First posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2019-03

CONDITIONS: Iron Status
Keywords: Iron Status; Iron deficiency; Cognition; Mood; Fatigue; Well-being; Women's Health
MeSH Terms: conditions — Iron Deficiencies; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood serum for serum ferritin analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Iron sufficient: Haemoglobin ≥120g/L Serum ferritin > 20μg/L
- Non-anaemic iron deficient: Haemoglobin ≥120g/L Serum ferritin ≤ 20μg/L
- Iron deficient anaemic: Haemoglobin <120g/L Serum ferritin ≤ 20μg/L
- Anaemic without iron deficiency: Haemoglobin <120g/L Serum ferritin > 20μg/L

SUMMARY:
Iron deficiency is the most prevalent nutritional deficiency worldwide with one in four estimated to be affected by iron deficiency anaemia. Women of reproductive age are at greatest risk for iron deficiency and anaemia due to iron losses during menstruation and childbirth as well as the increased need for iron throughout pregnancy. However, iron deficiency without anaemia is at least twice as common as iron deficiency anaemia with females aged 11-49 at the biggest risk of all. Despite this, it is commonly left undiagnosed. Those who are iron deficient non-anaemic can still suffer from the same common consequences of iron deficiency anaemia; these include unexplained fatigue, mood changes and decreased cognitive performance. Previous studies have found a significant relationship between iron status and cognitive performance in anaemic women. However, studies assessing cognition, mood and fatigue in women of varying iron status including those who are iron deficient nonanaemic are lacking. The most recent observational study of this kind found that better iron status was associated with better sustained attention but worse working memory. However, iron deficient anaemic females were not included in this observation. This study will extend upon this in order to determine any differences between non-anaemic iron deficiency and iron deficiency anaemia. The aims of this study are to improve knowledge concerning women's health and to determine whether there is a relationship between iron status, cognitive performance, subjective mood and fatigue in women of reproductive age (18-49 years).

DETAILED DESCRIPTION:
Each participant will be required to attend the laboratory on two occasions. The first is comprised of a screening/training visit, which will take place in the afternoon for approximately 2.5 hours. This will also be between days 21-28/the week before onset of their menstrual cycle. If they do not have menstrual bleeds then this appointment can be any afternoon. This will comprise: briefing of requirements of the study; obtaining of informed consent; confirmation of eligibility to take part, including collection of demographic data and health screening, and training on the cognitive and mood measures. The training session will follow standard operating procedures to decrease the chance of learning effects during main trials. Extra training will be given where necessary.

Participants will be required to complete questionnaires based upon food frequency, caffeine consumption and to estimate the number of hours of exercise completed on a weekly basis. A menstrual cycle questionnaire will also be completed to estimate menstrual blood loss and so that participants attend their testing visit during days 7-14 of their cycle. If participants do not have a menstrual cycle due to contraceptive methods, then appointments will be approximately two weeks apart.

A finger-prick and venous blood sample will be collected from participants, which will be analysed for iron status. Those whose haemoglobin levels are <120g/L will be advised to seek advice from their GP.

For the testing visit, participants will be asked to fast for 12 hours prior to the visit, avoiding intake of all food and drink with the exception of water. They will also be asked to avoid alcohol and refrain from intake of 'over the counter' medication for 24 hours. Participants will arrive at the laboratory at a designated time in the morning. The following procedures will take place prior to cognitive and mood testing:

* Review of continued conformity to eligibility criteria
* Adverse event and concomitant medication assessment
* Ensure that participant is in good health

Participants will then complete the baseline cognitive and mood assessments.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Female
* Aged 18-49 (inclusive)
* Have a BMI of between 18.5-40
* Have an English bank account (required for payment)

Exclusion Criteria:

* Aged under 18 or over 49
* BMI lower than 18.5 or higher than 40
* Pre-existing medical condition/illness with some exceptions - please check with researcher
* Blood disorders (excluding anaemia) or any known active infections
* Current or past breast cancer diagnosis and/or mastectomy
* Smoking or use of any nicotine replacement products e.g. vaping, gum, patches
* Pregnant, trying to get pregnant or breast feeding
* Currently taking any prescription medication with some exceptions - please check with researcher
* Regular use of dietary/herbal supplements within the last month (defined as more than 3 consecutive days or 4 days in total)
* Use of iron supplements within the past 4 months
* Have donated more than 300ml of blood in the past 3 months
* History of significant head trauma or suffer from frequent migraines that require medication (more than or equal to one per month)
* Learning difficulties, dyslexia, or colour blindness
* Visual impairment that cannot be corrected with glasses or contact lenses
* Currently taking part in any other clinical or nutritional intervention studies or have in the past 4 weeks
* Any health condition that would prevent fulfillment of the study requirements

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Must be female at birth
Study Population: Females aged 18-49 who meet the inclusion criteria who are based in Newcastle-upon-Tyne, United Kingdom and the residing North-East area.
Sampling Method: Non-Probability Sample
Enrollment: 379 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2019-04-03 (Actual)

PRIMARY OUTCOMES:
Speed of attention | Baseline measure
  An overall score for Speed of attention will be derived by calculating the average score from 3 separate standardised task outcomes (ZChoice reaction time correct reaction time + ZRapid visual information processing correct reaction time + ZDigit vigilance correct reaction time) /3
Subjective fatigue | Baseline measure
  Subjective fatigue will be derived from the total score of the Piper Fatigue Scale. Scores range from 1 to 10. Higher scores are indicative of greater fatigue.

SECONDARY OUTCOMES:
Episodic memory | Baseline measure
  An overall score for episodic memory will be derived by calculating the average score from 4 separate standardised task outcomes (Zimmediate word recall accuracy + Zdelayed word recall accuracy + Zword recognition accuracy + Zpicture recognition accuracy)/4
Speed of memory | Baseline measure
  An overall score for speed of memory will be derived by calculating the average score from 2 separate standardised task outcomes (Zpicture recognition correct reaction time + Zword recognition correct reaction time)/2
Accuracy of attention | Baseline measure
  An overall score for accuracy of attention will be derived by calculating the average score from 3 separate standardised task outcomes (ZChoice reaction time accuracy + ZZRapid visual information processing accuracy + ZZDigit Vigilance accuracy)/3
Executive function | Baseline measure
  An overall score for executive function will be derived by calculating the average score from 5 separate standardised task outcomes (Znumeric working memory accuracy + ZZserial 3 subtractions accuracy + ZZserial 7 subtractions accuracy + ZStroop accuracy - ZPeg and Ball errors)/5
Speed of executive function | Baseline measure
  An overall score for speed of executive function will be derived by calculating the average score from 3 separate standardised task outcomes (Znumeric working memory correct reaction time + Zstroop correct reaction time + ZPeg and Ball overall reaction time)/3
Computerised Location learning Task | Baseline measure
  An overall score is calculated utilising the total displacement over the 5 learning trials to create a total learning index score. Scores range from 0 to 1.
Subjective overall mood disturbance | Baseline measure
  Subjective mood disturbance is derived from the overall score of the Profile of Mood States questionnaire. Higher scores indicate a greater degree of overall mood disturbance.
Subjective sleep quality | Baseline measure
  Subjective sleep quality is derived from the overall score of the Sleep Condition Indicator. Total scores ranged from 0 to 32. Higher scores are indicative of greater subjective sleep quality.
Subjective stress | Baseline measure
  Subjective stress is derived from the overall score of the Perceived Stress Scale. Higher scores are indicative of greater subjective stress
Health Outcomes | Baseline measure
  Subjective health outcomes are derived from the SF-12. Scores range from 0 to 100. Higher scores are indicative of better self-reported health.
Subjective alertness | Baseline measure
  Subjective alertness will be derived from an Alertness visual analogue scale presented following cognitive task performance. Scores range from 0 to 100. Higher scores are indicative of greater feelings of alertness.
Subjective mental fatigue | Baseline measure
  Subjective mental fatigue will be derived from a Mental Fatigue visual analogue scale presented following cognitive task performance. Scores range from 0 to 100. Higher scores are indicative of greater feelings of mental fatigue.
Global Accuracy | Baseline measure
  An overall score for global accuracy will be derived by calculating the average score from 13 separate standardised outcomes (ZChoice reaction time accuracy + ZZRapid visual information processing accuracy + ZNumeric working memory accuracy + ZZDigit Vigilance accuracy + ZStroop accuracy - ZPeg and Ball Errors + ZZSerial 3 subtractions accuracy + ZZSSerial 7 subtractions accuracy + ZPicture recognition accuracy + ZWord recognition accuracy + ZImmediate word recall accuracy + ZDelayed word recall accuracy + ZZComputerised location learning accuracy)/13
Global Speed | Baseline measure
  An overall score for global speed will be derived by calculating the average score from 8 separate standardised outcomes (ZChoice reaction time correct reaction time + ZNumeric working memory correct reaction time + ZDigit vigilance correct reaction time + ZZPeg and Ball overall reaction time + ZStroop correct reaction time + ZPicture recognition correct reaction time + ZWord recognition correct reaction time + ZRapid visual information correct reaction time) /8

CONTACTS AND LOCATIONS:
Locations (1):
- Brain, Performance & Nutrition Research Centre, Northumbria University, Newcastle upon Tyne, United Kingdom

REFERENCES:
- [Background] Scott SP, Murray-Kolb LE. Iron Status Is Associated with Performance on Executive Functioning Tasks in Nonanemic Young Women. J Nutr. 2016 Jan;146(1):30-7. doi: 10.3945/jn.115.223586. Epub 2015 Dec 9. PMID 26661838
- [Background] Murray-Kolb LE, Beard JL. Iron treatment normalizes cognitive functioning in young women. Am J Clin Nutr. 2007 Mar;85(3):778-87. doi: 10.1093/ajcn/85.3.778. PMID 17344500
- [Background] Blanton CA, Green MW, Kretsch MJ. Body iron is associated with cognitive executive planning function in college women. Br J Nutr. 2013 Mar 14;109(5):906-13. doi: 10.1017/S0007114512002620. Epub 2012 Jun 7. PMID 22676919
- [Background] Fordy J, Benton D. Does low iron status influence psychological functioning? Journal of Human Nutrition and Dietetics 115: 167-183, 1994.